CLINICAL TRIAL: NCT04327310
Title: A Phase 1, 3 Part, Randomized, Placebo Controlled, Ascending Dose Study to Assess Safety, Tolerability, and Pharmacokinetics of Single Intravenous Doses of Meplazumab and to Assess Its Antimalarial Activity Against Plasmodium Falciparum in a Malaria Challenge Model in Healthy Subjects
Brief Title: Clinical Study of Meplazumab to Treat With Malaria
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The same drug has completed the phase I and II clinical trials for COVID-19
Sponsor: Jiangsu Pacific Meinuoke Bio Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMZ201501
Record Dates: First submitted 2020-03-24; First posted 2020-03-31 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-01

CONDITIONS: Malaria (Plasmodium Falciparum)
MeSH Terms: conditions — Malaria, Falciparum | interventions — meplazumab; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Meplazumab (Experimental): The vial of meplazumab will be reconstituted with 1 mL of water for injection. The required amount of drug solution will be withdrawn and added to 100 mL sterile normal saline (0.9%) for IV infusion. A single dose of meplazumab will be infused over 60 minutes at a constant rate using an infusion pump.
  Interventions: Drug: Meplazumab for Injection
- Placebo (Placebo Comparator): 100ml placebo will be infused over 60 minutes at a constant rate using an infusion pump, single time.
  Interventions: Drug: Sterile normal saline (0.9%)

INTERVENTIONS:
Drug: Meplazumab for Injection — humanized mAb against CD147
  Other Names: Meplazumab
  Arms: Meplazumab
Drug: Sterile normal saline (0.9%) — Sterile normal saline (0.9%)
  Arms: Placebo

SUMMARY:
This Phase 1 study will be conducted to explore the dose regimen in humans and to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and toxicological effects of meplazumab in healthy subjects, thus providing a new macromolecule antibody drug for the prevention and treatment of P. falciparum infection.

DETAILED DESCRIPTION:
2.1 Study Rationale.

This Phase 1 study will be conducted to explore the dose regimen in humans and to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and toxicological effects of meplazumab in healthy subjects, thus providing a new macromolecule antibody drug for the prevention and treatment of P. falciparum infection.

2.2 Background.

Malaria is a mosquito borne infectious disease that manifests as acute fever. Malaria is caused by Plasmodium spp., a parasite which is transmitted to humans by the bite of an infected female Anopheles mosquito (malaria vector).1 When the infected mosquito bites a human, Plasmodium sporozoites in the mosquito's saliva enter the bloodstream and migrate to the liver where they reproduce within hepatocytes. This stage is known as the exoerythrocytic phase.2 Multiplying merozoites reproduce to form schizonts, which contain several thousand merozoites. Mature schizonts rupture to release merozoites into the blood where they invade erythrocytes,3 hence initiating the merozoites reproduction in the erythrocytic phase.2 Malaria may develop into severe or even fatal disease if not treated in time. Five species of Plasmodium infect humans, including Plasmodium falciparum (P. falciparum), P. vivax, P. ovale, P. malariae, and P. knowlesi.4 Among these, P. falciparum and P. vivax are the most common species, with the former as the most dangerous one which has a high morbidity and may result in rapid progression and high mortality.

Current methods toward malaria elimination usually involve the combination of prevention and treatment. Early diagnosis and treatment can mitigate disease progression and reduce deaths. Artemisinin based combination therapies are currently recommended by the World Health Organization for treatment of malaria. Antimalarial drugs mainly include drugs to eliminate Plasmodium during the erythrocytic phase or during the exoerythrocytic phase.

From the 1950s, falciparum malaria has progressively developed resistance to all antimalarials marketed including chloroquine, sulfadoxine pyrimethamine, etc leading to ineffective malaria control. Plasmodium spp. Have recently developed resistance to the current frontline drugs, artemisinin combination therapy. Therefore, new antimalarial therapies and drugs are urgently needed to combat drug resistance of Plasmodium.

2.2.1 Meplazumab, a Humanized Anti-CD147 IgG2 Monoclonal Antibody

Meplazumab (Ketantin®) is a lyophilized powder for injection of small volume. The main active ingredient of the product, meplazumab, is a humanized immunoglobulin (Ig) G2 monoclonal antibody, consisting of the complementary-determining regions of anti CD147 murine antibody and the human framework region. It acts as an erythrocytic stage-macromolecular antibody drug that has the potential to mediate both treatment and prophylaxis of falciparum malaria.

2.2.2 Preclinical Data

Preclinical studies and pharmacological studies have indicated that meplazumab for intravenous (IV) injection is safe and effective with well controlled quality. The nonclinical studies of meplazumab include pharmacology, PD, PK, and toxicology studies. Refer to Section 4 of the current IB for meplazumab for further details.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent as described in Appendix 2, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol, prior to any study-specific procedures.
* Men and women aged 18 to 55 years (inclusive), with suitable veins for cannulation or repeated venipuncture.
* Total body weight ≥50 kg, and a body mass index between 18 to 32 kg/m2, inclusive.
* Female subjects are eligible to participate if they have a negative pregnancy test at the Screening Visit and on admission to the study center, not lactating
* Male subjects with female partners of childbearing potential must agree to use contraception as detailed in Appendix 7 of this protocol from the time of informed consent until at least 3 months after dosing with the investigational product. Male subjects with female partners that are surgically sterile, or male subjects who have undergone sterilization and have had testing to confirm the success of the sterilization, may also be included.
* Male subjects must not donate sperm from the day of dosing until at least 3 months after dosing with the investigational product.
* Medically healthy with clinically insignificant screening results based on a comprehensive medical history and physical examination as judged by the Principal Investigator.
* Has to agree to abstain from alcohol intake 48 hours before administration of the study treatment and inoculation with P. falciparum, and during the confinement period of the study.
* Able to be compliant with the protocol and attend all scheduled visits.

Exclusion Criteria:

* Previously treated with study treatment in the present study.
* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Any known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product.
* History of splenectomy.
* Subjects with history of schizophrenia, bi-polar disease, psychoses, disorders requiring lithium, attempted or planned suicide, or any other severe (disabling) chronic psychiatric diagnosis.
* Subjects who have been hospitalized within 5 years prior to enrollment for either a psychiatric illness or due to danger to self or others.
* History of an episode of minor depression that required at least 6 months of pharmacological therapy and/or psychotherapy within the last 5 years; or any episode of major depression.
* Presence of clinically significant infectious disease or fever (eg, sublingual temperature ≥38.5°C) within 5 days prior to study treatment administration (Parts A and C) or inoculation with the malaria challenge agent (Part B).
* Hematology, biochemistry, or urinalysis results at Screening or at Day -1 (Parts A and C) or between Day -11 to -9 (Part B) that are outside of Sponsor-approved clinically acceptable laboratory ranges (Appendix 4), or are considered clinically significant by the Investigator. One repeat is permitted at Screening.
* Any positive result at Screening for hepatitis B surface antigen, anti-hepatitis B core antibodies, rapid plasma reagin, anti-hepatitis C virus antibody, and anti-human immunodeficiency virus 1 and 2 antibodies.
* Symptomatic postural hypotension at Screening (confirmed on 2 consecutive readings), irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 2 to 3 minutes when changing from supine to standing position.
* Abnormal vital signs at Screening (supine and standing) and on Day 1 (Parts A and C) or pre-inoculation on Day 8 (Part B) (supine), defined as any of the following:

  1. Systolic blood pressure <90 or >140 mmHg.
  2. Diastolic blood pressure <40 or >90 mmHg.
  3. Pulse rate <40 or >100 bpm.
* Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG, and any clinically important abnormalities in the 12 lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval changes.
* Prolonged Fridericia QT correction formula (QTcF) (>450 msec for males and >470 msec for females), prolonged Bazett's QT correction formula (QTcB) (>450 msec for males and >470 msec for females), or PR interval >210 msec (both males and females), or shortened QTcF <340 msec or family history of long QT syndrome at the Screening Visit and on Day 1 (Parts A and C) or pre-inoculation on Day -8 (Part B).
* Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss >500 mL or blood transfusion during the 3 months prior to the Screening Visit. For Parts B and C, subjects who have ever received a blood transfusion will be excluded.
* Current smokers (tobacco use of >5 cigarettes or equivalent per day), or those unable to stop smoking during confinement.
* History of alcohol abuse or excessive intake of alcohol defined as an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to 12 g alcohol = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80-proof distilled spirits.
* History of drug habituation, or any prior intravenous usage of an illicit substance.
* Positive urine drug and alcohol breath test at Screening or on admission to the study center prior to the administration of investigational product (Day -1 for Parts A and C and Day 1 for Part B)/inoculation with malaria challenge agent (Day -8 for Part B and Day 3 for Part C). Positive for any drug listed in Appendix 4 in the urine drug screen, unless there is an explanation acceptable to an Investigator (eg, the subject has stated in advance that they consumed a prescription or over-the-counter product which contained the detected drug) and/or the subject has a negative urine drug screen on retest by the pathology laboratory. Any subject testing positive for acetaminophen (paracetamol) at Screening and/or inoculation day may still be eligible for study participation, at the Investigator's discretion.
* Excessive intake of caffeine-containing drinks or food, eg, coffee, tea, chocolate, Red Bull, or cola (more than 400 mg of caffeine per day, equivalent to >4 cups of coffee per day) for 48 hours before the start of dosing or inoculation with malaria challenge agent.
* Ingestion of any poppy seeds within 24 hours prior to each Drug Abuse Screening (Screening Visit [all Parts], Day 1 [Part A and Part C], Day -8 and Day 1 [Part B], and Day 3 [Part C]). Subjects will be advised by phone not to consume any poppy seeds in this time period.
* Any history or presence of diagnosed (by an allergist/immunologist) or treated (by a physician) food or known drug allergies, or history of anaphylaxis or other severe allergic reactions including face, mouth, or throat swelling or any difficulty breathing. Subjects with seasonal allergies/hay fever or allergy to animals or house dust mite that are untreated and asymptomatic at the time of dosing can be enrolled in the study.
* Use of any prescribed or nonprescribed medication including antacids, analgesics, herbal preparations, or vitamins (other than paracetamol/acetaminophen [<4 g per day], ibuprofen [<1.2 g per day], or routine vitamins [megadose intake of 20 to 600 times the recommended daily dose is prohibited]) within 2 weeks prior to the first administration of investigational product or 5 times the medication's half life, whichever is longer. Limited use of other non prescription medications or dietary supplements, not believed to affect subject safety or the overall results of the study, may be permitted a case-by-case basis following discussion with the Investigator and approval of the Sponsor. Hormone replacement therapy is allowed.
* Any vaccination within the last 28 days.
* Any recent (<6 weeks) or current systemic therapy with an antibiotic or drug with potential antimalarial activity (eg, chloroquine, piperaquine phosphate, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, doxycycline etc.).
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within 3 months of the administration of investigational product in this study. The period of exclusion begins 3 months after dosing (or greater than 5 times half life) or 1 month after the last visit, whichever is the longest. Note: Subjects consented and screened, but not dosed in this study or a previous Phase I study, are not excluded.
* Involvement in the planning and/or conduct of the study (applies to the Sponsor, contract research organizations, and study center staff, etc.).
* Subjects who are unlikely to co operate with the requirements of the study.
* Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Presence of Anti-antibodies | Time Frame: 71±3 days (throughout the study period)
  collection of blood samples for immunogenicity assessments，using vadiation Anti-body testing assay to test the presence of anti-antibodies
Adverse events / serious adverse events | 43±3 days (from first dose to end of study)
  Recording of adverse events / serious adverse events throughout the study period

SECONDARY OUTCOMES:
The area under the plasma drug concentration-time curve (AUC) | 43±3 days (from first dose to end of study)
  Meplazumab serum concentration
Maximum Plasma Concentration | 43±3 days (from first dose to end of study)
Time to Maximum Plasma Concentration | 43±3 days (from first dose to end of study)
Area under the serum concentration-time curve from time zero extrapolated to infinity | 43±3 days (from first dose to end of study)
  Calculated by linear up/log down trapezoidal summation
Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration | 43±3 days (from first dose to end of study)
  Calculated by linear up/log down trapezoidal summation
Terminal half-life | 43±3 days (from first dose to end of study)
  A minimum of 3 points will be used for estimation
Systemic clearance | 43±3 days (from first dose to end of study)
Volume of distribution | 43±3 days (from first dose to end of study)
Volume of distribution at steady state | 43±3 days (from first dose to end of study)